CLINICAL TRIAL: NCT01846702
Title: A Single-Dose, Dose-Escalation Study to Determine the Safety, Tolerability, and Pharmacokinetics of LY3084077 in Healthy Subjects
Brief Title: A Study of LY3084077 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14530; I6P-MC-FMRA (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of placebo matching LY3084077 administered subcutaneously (SC).
  Interventions: Drug: Placebo
- LY3084077 (Experimental): Single escalating doses (1 mg up to 300 mg) of LY3084077 administered SC.
  Interventions: Drug: LY3084077

INTERVENTIONS:
Drug: Placebo — Given as a SC injection.
  Arms: Placebo
Drug: LY3084077 — Given as a SC injection.
  Arms: LY3084077

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY3084077 in healthy participants. The study will also investigate how much of the study drug gets into the blood stream and how long it takes the body to get rid of it. Information about any side effects that may occur will also be collected. The study is expected to last approximately 8 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have normal blood pressure
* Must be a healthy male or female who cannot become pregnant
* Have a body mass index (BMI) of 18.5 to 40.0 kg/m^2, inclusive, at screening

Exclusion Criteria:

* Have known allergies to fibroblast growth factor-21 (FGF21) analogues, glucagon-like peptide-1 (GLP1), GLP1-analogues or other related compounds
* Have previous exposure to FGF21 analogues or GLP1 analogues
* Have received live vaccine(s) within 1 month of screening, or intend to during the study
* Have previously completed or withdrawn from this study
* Have or used to have health problems or laboratory test results or electrocardiogram (ECG) readings that in the opinion of the doctor, could make it unsafe to participate, or interfere with understanding the results of the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Have problems with the immune system, due to a disease or treatment
* Have a personal or family history of medullary thyroid carcinoma (MTC) or have multiple endocrine neoplasia syndrome type 2
* Have a history of pancreatitis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Cohort 1: Single dose of placebo matching LY3084077 administered subcutaneously (SC).
- LY3084077 Cohort 2: 1 mg single dose of LY3084077 administered SC.
- LY3084077 Cohort 3: 3 mg single dose of LY3084077 administered SC.
- LY3084077 Cohort 4: 10 mg single dose of LY3084077 administered SC.
- LY3084077 Cohort 5: 30 mg single dose of LY3084077 administered SC.
- LY3084077 Cohort 6: 100 mg single dose of LY3084077 administered SC.
- LY3084077 Cohort 7: 150 mg single dose of LY3084077 administered SC
Period: Overall Study
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Started | 6 | 6 | 7 | 6 | 6 | 6 | 6
Received at Least 1 Dose of Study Drug | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- LY3084077 Cohort 4: 10 mg single dose of LY3074077 administered SC.
- LY3084077 Cohort 5: 30 mg single dose of LY3074077 administered SC.
- LY3084077 Cohort 6: 100 mg single dose of LY3074077 administered SC.
- LY3084077 Cohort 7: 150 mg single dose of LY3074077 administered SC.
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (14) | 30.7 (13.2) | 34.5 (11.2) | 32.7 (7.4) | 40.7 (12.6) | 30.5 (5.0) | 36.3 (4.8) | 34.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Male | 6 | 5 | 6 | 6 | 5 | 6 | 6 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 4 | 6 | 6 | 6 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: An SAE is an adverse event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Pre-dose, Up to Day 190
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Placebo Cohort 1: Single dose of placebo matching LY3084077 administered SC.
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 1 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Zero to Infinity (AUC[0-∞]) GLP1-Fc Domain of LY3084077
Time Frame: Day 1 and Day 29: Predose, 2,4,8,12,24,36,48,72,96,120,168,336 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (μg•hr/mL)
Groups:
- LY3084077 Cohort 3: 3mg single dose of LY3084077 administered SC.
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 2 | 5 | 4 | 6 | 6
microgram*hour/milliliter (μg•hr/mL) | NA (NA) — Cohort 1 was not calculable due to samples from placebo treated participants were not analyzed. | NA (NA) — Cohort 2 was not calculable due to concentration level was below quantification limits. | 8.74 (13) | 17.9 (42) | 61.8 (34) | 248 (221) | 249 (20)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) GLP1-Fc Domain of LY3084077
Time Frame: Day 1 and Day 29: Predose, 2,4,8,12,24,36,48,72,96,120,168,336 hours post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 6 | 6 | 6
microgram/milliliter (μg/mL) | NA (NA) — Cohort 1 was not calculable due to samples from placebo treated participants were not analyzed. | NA (NA) — Cohort 2 was not calculable due to concentration level was below quantification limits. | 0.0428 (53) | 0.0745 (24) | 0.188 (78) | 1.14 (79) | 1.23 (48)

4. Secondary Outcome: Pharmacodynamics (PD): Percent Change From Baseline in Fasting Triglycerides
Description: Percent change=(measure at time t-measure at baseline)/measure at baseline*100%). Least Square Means (LS means) were calculated using MMRM analysis adjusting for the random effect of participant, effect of baseline, and fixed categorical effects of treatment, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Up to Day 15
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting triglycerides data.
Measure: Least Squares Mean (Standard Deviation); unit: percent
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
percent | -23.7 (12.8) | -13.7 (12.8) | -35.3 (12.6) | -30.4 (12.6) | -23.8 (13.6) | -2.50 (14.2) | -43.7 (13.0)

5. Secondary Outcome: PD: Change From Baseline in Fasting Insulin
Description: LS means were calculated using MMRM analysis adjusting for the random effect of participant, effect of baseline, and fixed categorical effects of treatment, visit, and treatment-by-visit interaction.
Time Frame: Baseline, Up to Day 15
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting insulin data.
Measure: Least Squares Mean (Standard Error); unit: picomole/Liter (pmol/L)
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
picomole/Liter (pmol/L) | -24.0 (8.23) | -24.6 (8.55) | -21.4 (8.41) | 4.90 (8.26) | -28.4 (9.19) | -11.9 (8.29) | -26.6 (8.44)

6. Secondary Outcome: PD: Change From Baseline in Weight
Time Frame: Baseline, Up to Day 15
Population: Zero participants had weight measured and therefore change from baseline in weight was not calculable across all arms.
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: PD: Change From Baseline Up to Day 2 in Level of C-peptide AUC (Predose to 4 Hours) After a Standard Meal
Description: as for outcome 5
Time Frame: Baseline, Day 2
Population: All randomized participants who received at least one dose of study drug and had evaluable C-peptide AUC before and after a standard meal data.
Measure: Least Squares Mean (Standard Error); unit: picomole*hour/Liter (pmol*h/L)
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
picomole*hour/Liter (pmol*h/L) | -292 (579) | 310 (559) | -157 (579) | 1313 (564) | 372 (592) | -192 (564) | 973 (568)

8. Secondary Outcome: PD: Change From Baseline to Day 2 Incremental AUC Level of Blood Glucose (Predose to 6 Hours) After a Standard Meal
Description: as for outcome 5
Time Frame: Baseline, Day 2
Population: All randomized participants who received at least one dose of study drug and had evaluable incremental glucose AUC before and after a standard meal data.
Measure: Least Squares Mean (Standard Error); unit: millomole*hour/Liter (mmol*h/L)
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
millomole*hour/Liter (mmol*h/L) | -1.76 (1.16) | 0.758 (1.18) | -0.202 (1.14) | -0.350 (1.15) | -2.14 (1.13) | -1.79 (1.13) | -1.82 (1.15)

9. Secondary Outcome: PD: Change From Baseline to Day 2 in Fasting Glucagon
Description: as for outcome 5
Time Frame: Baseline, Up to Day 2
Population: All randomized participants who received at least one dose of study drug and have evaluable fasting glucagon data.
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
pmol/L | 3.17 (1.98) | 0.940 (1.96) | 2.38 (1.98) | -0.514 (1.95) | 4.15 (1.96) | 1.01 (1.99) | 1.52 (1.96)

10. Secondary Outcome: Number of Participants Developing Anti-LY3084077 Antibodies
Description: The number of participants with 1:4 baseline and postbaseline positive anti-LY3084077 antibody titers.
Time Frame: Pre-dose, Up to Day 190
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and postbaseline antibody titers.
Measure: Number; unit: participants
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
participants | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo Cohort 1 | LY3084077 Cohort 2 | LY3084077 Cohort 3 | LY3084077 Cohort 4 | LY3084077 Cohort 5 | LY3084077 Cohort 6 | LY3084077 Cohort 7
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/6 | 3/6 | 5/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=6) | LY3084077 Cohort 2 (N=6) | LY3084077 Cohort 3 (N=6) | LY3084077 Cohort 4 (N=6) | LY3084077 Cohort 5 (N=6) | LY3084077 Cohort 6 (N=6) | LY3084077 Cohort 7 (N=6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=6) | LY3084077 Cohort 2 (N=6) | LY3084077 Cohort 3 (N=6) | LY3084077 Cohort 4 (N=6) | LY3084077 Cohort 5 (N=6) | LY3084077 Cohort 6 (N=6) | LY3084077 Cohort 7 (N=6)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 3 (3) | 4 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No